CLINICAL TRIAL: NCT04520399
Title: Prediction of Violent Behavior in Patients With Schizophrenia by Multimodal Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20200498
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia; Violence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- violence
  Interventions: Other: none intervention
- non-violence
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — there is no intervention in this study

SUMMARY:
Patients with schizophrenia have a higher risk of committing violent crimes than the general population, and the relative risk of violence against others is four times higher than the general population. Violence is a major public health problem because it often leads to poor prognosis, readmission and stigma in patients with schizophrenia.

MRI studies on violent behavior in schizophrenia are relatively few. These studies have found that violence is primarily associated with dysfunction in the ventral prefrontal and temporal limbic systems. Structural MRI found that violent behavior in schizophrenia was associated with increased volume of white matter in caudate nucleus, left orbitofrontal gyrus and right orbitofrontal gyrus. However, the current research results in this field are uneven, the methods are not consistent, and there is a lack of breakthrough progress, which needs to be integrated and deepened urgently.

If the violent behavior of the patients with schizophrenia could be predicted by magnetic resonance imaging, it would be a revolutionary try. By doing so, the investigators can strengthen the treatment of these patients and reduce the occurrence of violence. Based on previous studies, the investigators believe that violent schizophrenics exhibit recognizable imaging characteristics under structural phase, resting state, negative emotional images and natural stimuli models. Anomalies in a particular mode may be subtle and difficult to identify, but when multiple different modes are integrated, a significant and characteristic set of imaging markers will be present. This study will use the multivariate model of machine learning method, detection brain activation patterns under different situations among patients with violence. The investigators are going to study imaging biomarkers, and try to predict the possibility of onset of violence among schizophrenia patients, thus reduce the risks of violence.

ELIGIBILITY:
Inclusion Criteria:

for violent group

1. Inpatient or out-patient treatment;
2. Junior high school education or above, eliminate mental retardation;
3. 18-60 years old;
4. Han, right-handed;
5. Meet the diagnostic criteria of ICD-10 schizophrenia;
6. Self-report and confirmed by family members that violence occurred at least 2 times in the recent six months;
7. In the recent half year, the revised Version of the weighted total score of The Explicit Attack Scale (MOAS) ≥4;
8. Exclude severe heart, liver, kidney, blood, digestive and nervous system diseases;
9. Willing to participate in this study and sign the informed consent. Inclusion criteria for non-violent patients

1) Schizophrenic patients treated in hospital or outpatient; 2) Junior high school education or above, eliminate mental retardation; 3) 18-60 years old; 4) Han, right-handed; 5) Meet the diagnostic criteria of ICD-10 schizophrenia; 6) Self-reported and confirmed by family members that no violence has occurred in the past six months; 7) within the past revisions explicit scale (MOAS) weighted total score ˂ 4 points; 8) Exclude severe heart, liver, kidney, blood, digestive and nervous system diseases; 9) Willing to participate in this study and sign the informed consent.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 200 schizophrenic patients were collected in Shanghai Mental Health Center. Through the assessment of violent behavior (MOAS scale + self-report), schizophrenic patients were divided into violent group and non-violent group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
MRI testing results | Sep.2022
  structural MRI data
resting state MRI data | Sep.2020
  functional connections between brain regions
functional MRI data | Sep.2020
  brain stimulation models while in a natural stimulus or watching affective pictures
Integrated data | Sep.2020
  integrated MRI data from machine learning method

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No